CLINICAL TRIAL: NCT00585039
Title: Comparison of Hospital Admission Rates and Plasma(s)-Albuterol Levels in Children Treated With Racemic Albuterol Versus Levalbuterol for Acute Asthma Exacerbations: A Randomized Double-Blind Clinical Trial
Brief Title: Albuterol Versus Xopenex in Treatment of Acute Asthma in the Emergency Department (ED)
Acronym: Xopenex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRC176
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Results first posted 2011-08-16 (Estimated); Last update posted 2026-02-10 (Actual); Status verified 2011-09

CONDITIONS: Asthma
Keywords: child; emergency department
MeSH Terms: conditions — Asthma; Emergencies | interventions — Levalbuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): levalbuterol nebulization
  Interventions: Drug: xopenex

INTERVENTIONS:
Drug: xopenex — will receive xopenex rather than albuterol to treat acute exacerbation
  Other Names: levalbuterol

SUMMARY:
The purpose of this study is to determine in a large, double-blind, randomized, prospective pediatric clinical trial whether the use of continuous levalbuterol (Xopenex) in addition to standard emergency department treatment for acute asthma exacerbations will improve the Forced Expiratory Volume in 1 sec (FEV 1) compared to the use of continuous racemic albuterol. The secondary objective is to correlate clinical (hospitalization rates and clinical asthma scores) with plasma levels of (S)-albuterol.

DETAILED DESCRIPTION:
Children between the ages of 6 and 17 years inclusive who have a history of asthma are eligible for enrollment if they present to the pediatric emergency department with a moderate to severe acute asthma exacerbation. All eligible children will be enrolled whenever there are study personnel available after obtaining informed written consent. Children less than 6 years of age will not be enrolled as levalbuterol has only been approved in children 6 years of age and greater. Children will also be excluded if their Forced Expiratory Volume in 1 sec (FEV 1) is > 70% predicted (see below); they have a history of a chronic lung disease (e.g. cystic fibrosis), noncorrected congenital heart disease, suspected intrathoracic foreign body, need immediate resuscitation or are pregnant.

Eligible patients will be identified by research assistants and the attending ED physician will be notified. The attending ED physician will make the final decision regarding severity based on their physical exam and spirometry (FEV 1) results. The FEV 1 value will be recorded and calculated as a percentage of their predicted based on standardized height and weight charts. All spirometry will be performed by licensed respiratory therapists or research assistants trained in the use of the spirometer. An FEV 1 of 50% to 70% predicted will be considered a moderate exacerbation and if less than 50% predicted, severe.

As the children being enrolled are having significant asthma exacerbations there will be no delay in their treatment. If the consent process can not be carried within the first 15 minutes upon arrival to the ED they will receive a standard dose of albuterol as per our standing ED orders.

A computer generated table of random numbers will be used to assign children to treatment group. A locked area in the ED will contain numbered plastic bags each containing either 15 mg of racemic albuterol or 7.5 mg of levalbuterol. Since we are only enrolling children ≥ 6 years of age they should all weigh > 20 kg and therefore will receive 7.5 mg of racemic albuterol (0.5%, 2.5mg/0.5 ml Nephron Pharmaceuticals) in normal saline (total volume = 20 ml) nebulized over one hour if assigned to the albuterol group (i.e. the equivalent of 2.5 mg every 20 minutes for 3 doses). If they are between 6 and 11 years of age they will receive 1.89 mg levalbuterol and if ≥ 12 years of age 3.75 mg of levalbuterol in the same volume of normal saline. This would be the equivalent of giving 3 treatments every 20 minutes for one hour. Both study medications will be identical in odor and appearance. All children will receive 2 mg/kg of methylprednisolone up to a maximum dose of 60 mg orally within the first 20 minutes of treatment. All children will also receive two unit doses of ipratropium bromide (1000 mcg) in the first hour of nebulization therapy as this is standard of care.

Spirometry will be performed at baseline and after each hour of bronchodilator treatment until the child is discharged home or is admitted to an in-patient unit. Patient disposition from the ED depends on their response to treatment. The ultimate decision to admit or discharge will be at the attendings discretion. However, if the child is able to perform good loops on spirometry then FEV1 may be used to guide the decision. An FEV 1 ≥ 70% predicted will likely mean discharge to home with appropriate instructions. Children will be observed for 60 minutes after their last bronchodilator treatment to ensure that they maintain their response. Children will be admitted to the PICU if their FEV 1 < 50% or if they require inhaled bronchodilators more than hourly. If the child's FEV 1 is ≥ 50% but < 70% or if they are still experiencing moderate symptoms they are likely to be admitted to the floor but further treatment in the ED may allow sufficient improvement for discharge. If after a further treatment period of one hour their FEV1 is > 70% they will be discharged home. If it is < 70% they will be admitted. Once disposition has been decided the study is concluded for that patient except for telephone follow-up if the child was discharged home.

All children discharged home will be called 30 days after their ED assessment. This call will determine if the child had any further unscheduled ED or office visits for the same asthma exacerbation.

Data to be collected include the child's age, weight, height, gender, ethnicity, medication use at home, asthma history, asthma scores, peak flows, disposition from ED, adverse effects, and serum levels of the albuterol isomers (see data collection sheet attached).

Blood will be drawn at baseline. The serum level for albuterol enantiomers requires 7 ml of blood and will only be drawn once. Children can elect to be in just the RCT of the two medications or to take part in both parts of the study. Blood samples will be sent to the lab, spun down and frozen. The samples will be stored there until the study is completed and then shipped to an outside lab for measurement of plasma levels of (S) and (R) albuterol. These plasma levels will only be reviewed after patient disposition has already been decided as they are not clinically relevant to their acute management at this time.

There will be dedicated research personal in the ED 16 hours a day for the sole purpose of identifying study candidates and ensuring all procedures are followed according to the protocol. This is to ensure continuity through the study process including placement of the consent in the medical record. Since spirometry is an objective test it also allows for shift changes without the need to worry about a different individual measuring the FEV1. Despite this all ED staff (physicians, fellows, nurses, technicians) will be informed and educated on the purpose, protocol and procedures to be used in the study at regularly scheduled staff meetings.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between the ages of 6 and 17
* Has previously been diagnosed with asthma by any physician
* Has presented to the ED with an asthma exacerbation judged by a physician to be of a moderate or severe degree

Exclusion Criteria:

* Requires immediate resuscitation (attending physician)
* Is pregnant and/or breast feeding
* If possibly pregnant, negative pregnancy test attached
* Has chronic lung diseases (i.e. cystic fibrosis)
* Has an uncorrected congenital heart diseaseHas a suspected foreign body aspiration
* Is allergic to albuterol and/or levalbuterol (Xopenex)
* Has an initial FEV 1>70% predicted

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2005-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bulloch, MD, Principal Investigator — Phoenix Children's Hospital
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children 6 to 17 years who presented to ED with asthma exacerbation of moderate to severe nature.
Pre-assignment Details: 2 children were excluded from levalbuterol group after enrollment, 1 because the study medication spilled and another because they had received the medication outside protocol timeline. All other enrolled patients completed study.
Groups:
- Levalbuterol (Xopenex): Patients who received 3.75 mg levalbuterol nebulization at baseline and could be repeated at 60 minutes
- Albuterol: patients who received 7.5 mg albuterol nebulization at baseline and could be repeated at 60 minutes
Period: Overall Study
Arm/Group | Levalbuterol (Xopenex) | Albuterol
Started | 57 | 44
Completed | 55 | 44
Not Completed | 2 | 0
Not completed — medication spilled | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levalbuterol (Xopenex) | Albuterol | Total
Number analyzed (Participants) | 57 | 44 | 202
Age, Categorical [Count of Participants; unit: Participants]
  number analyzed (Participants) | 57 | 44 | 101
  <=18 years | 57 | 44 | 101
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  number analyzed (Participants) | 57 | 44 | 101
  Female | 39 | 33 | 72
  Male | 18 | 11 | 29
Region of Enrollment [Number; unit: participants]
  United States: number analyzed (Participants) | 57 | 44 | 101
  United States | 57 | 44 | 101

OUTCOME MEASURES:

1. Primary Outcome: Change in Forced Expiratory Volume in 1 Sec (FEV1) Measured in L/Sec
Time Frame: Baseline and 4 hours
Population: Enrollment period ended prior to final goal sample size. ITT.
Measure: Mean (95% Confidence Interval); unit: L/sec
Arm/Group | Levalbuterol (Xopenex) | Albuterol
Number analyzed (Participants) | 55 | 44
L/sec | 19.8 [14.4 to 67] | 55.2 [28 to 75.7]

2. Secondary Outcome: Clinical Asthma Score (CAS)
Description: Change in clinical asthma score while in ED. 15 point clinical asthma score. Score ranges from 5 (no to mild respiratory distress) to a maximum of 15 (severe respiratory distress).
Time Frame: 4 hours
Population: analysis per protocol
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Levalbuterol | Albuterol
Number analyzed (Participants) | 55 | 44
units on a scale | 1.7 [0 to 2.9] | 3.0 [1.2 to 3.9]

ADVERSE EVENTS:
Arm/Group | Levalbuterol (Xopenex) | Albuterol
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/44
Other Adverse Events (participants affected / at risk) | 0/55 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No